CLINICAL TRIAL: NCT07296744
Title: Pivotal Randomized Study of the SUpira System in Patients Undergoing High-Risk Percutaneous COronaRy InTervention (HRPCI)
Brief Title: Pivotal Study of the SUpira System in Patients Undergoing High-Risk Percutaneous COronaRy InTervention (HRPCI)
Acronym: SUPPORT II
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Supira Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-10004
Record Dates: First submitted 2025-12-18; First posted 2025-12-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Disease; High Risk Percutaneous Coronary Intervention; Interventional Cardiology; Mechanical Circulatory Support
Keywords: Percutaneous ventricular assist device; Supira System; Mechanical Circulatory Support; US Pivotal
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: This is a prospective, multicenter, open label, randomized controlled trial (RCT). Subjects undergoing HRPCI will be randomized (1:1)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Supira System (Experimental): Subjects receiving the Supira System
  Interventions: Device: The Supira System
- Impella (Active Comparator): Subjects receiving the Impella
  Interventions: Device: Impella

INTERVENTIONS:
Device: The Supira System — The Supira System is a temporary (≤ 4 hours) ventricular support device indicated for use during elective or urgent HRPCI performed in hemodynamically stable patients with severe coronary artery disease when a heart team has determined HRPCI is the appropriate therapeutic option.
  Arms: Supira System
Device: Impella — The current commercially available Impella CP with SmartAssist Catheter is indicated for providing temporary (≤ 6 hours) ventricular support during elective or urgent high risk percutaneous coronary i
  Arms: Impella

SUMMARY:
The objective of this study is to assess the safety and efficacy of the Supira System in providing temporary cardiovascular hemodynamic support in patients undergoing HRPCI. Eligible patients will be randomized to undergo HRPCI with either the Supira System (investigational device) or the commercially available Impella systems (comparator device).

DETAILED DESCRIPTION:
The Supira System is a minimally invasive percutaneous ventricular assist device (pVAD) that is intended to provide temporary hemodynamic support (≤ 4 hours) to patients undergoing HRPCI. The Supira Catheter is inserted percutaneously through the femoral artery, across the aortic valve, and into the left ventricle under fluoroscopic guidance, with the pump outlet remaining in the ascending aorta. The pump portion of the Catheter compresses during insertion in the Introducer Sheath and re-expands during use. It actively unloads the left ventricle by pumping blood from the ventricle into the ascending aorta and systemic circulation.

ELIGIBILITY:
Inclusion Criteria:

* Hemodynamically stable and will undergo elective or urgent (not emergent) HRPCI, where hemodynamic support is deemed necessary, as determined by the institutional Heart Team
* Informed consent granted by the subject or legally authorized representative

Exclusion Criteria:

* Cardiogenic shock or acutely decompensated pre-existing chronic heart failure
* Stroke within 6 months of the index procedure, or any prior stroke with permanent neurologic deficit
* Left ventricular thrombus
* Aortic and iliofemoral anatomical conditions that preclude safe delivery and placement of the investigational device or the comparator device
* Ongoing renal replacement therapy with dialysis
* Presence of decompensated liver disease; severe liver dysfunction
* Infection of the proposed procedural access site or active infection
* Known hypersensitivity to intravenous contrast agents that cannot be adequately pre-medicated or known hypersensitivity to heparin, aspirin, adenosine diphosphate (ADP) receptor inhibitors, or nitinol
* Any condition, coagulopathy, planned procedure or contraindication that requires discontinuation of antiplatelet and/or anticoagulant therapy within 90 days of the index procedure
* Breastfeeding or pregnant or planning to become pregnant within 90 days of the HRPCI procedure
* Currently participating in active follow-up phase of another clinical study of an investigational drug or device or planning to enroll in such a study within 90 days of the HRPCI procedure
* Other medical, social, or psychological problems that, in the opinion of the Investigator, compromises the subject's ability to provide written informed consent and/or to comply with study procedures
* Considered to be part of a vulnerable population per the investigator's assessment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Composite Safety and Efficacy Outcomes | 30 days
  * All-cause death
  * Myocardial infarction
  * Stroke or transient ischemic attack
  * Major bleeding
  * Major access site-related vascular complications
  * Acute Kidney Injury
  * Unplanned repeat revascularization
  * Sustained hypotensiona during mechanical circulatory support
  * Arrythmia requiring cardioversion during pump use

SECONDARY OUTCOMES:
Secondary Outcome Measures | 30 and 90 days
  Individual rates of the following outcomes:
  * All-cause death
  * MI
  * Stroke or TIA
  * Major bleeding
  * Major access site-related vascular complications
  * AKI
  * Unplanned repeat vascularization
  * Cardiovascular re-hospitalization
  * Ventricular arrhythmia requiring cardioversion
  * Major cardiac structural complications
  * Major Hemolysis

IPD SHARING:
Plan to Share IPD: No